CLINICAL TRIAL: NCT01159717
Title: Complex Cystic Renal Lesions: Evaluation of Computed Tomography Findings With Contrast Enhanced Ultrasound in Terms of the Bosniak Classification System.
Brief Title: CT Versus CEUS Findings of Complex Cystic Renal Lesions
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Dr. Joachim Hohmann, Department of Radiology
Other Study IDs: EK 129/09
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Kidney Neoplasms; Computed Tomography; Ultrasonography; Contrast Media
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective comparison of complex cystic renal lesions which are found with computed tomography (CT) and were controlled with contrast enhanced ultrasound (CEUS).

DETAILED DESCRIPTION:
All subjects receive an contrast enhanced CT due to different clinical indications. When a complex cystic renal lesion is found an evaluation with CEUS is performed. The CEUS protocol included a native baseline examination of both kidneys. After a bolus injection of 1.5 ml SonoVue (Bracco, Milano, Italy) an examination of the affected kidneys is performed over a time period of at least three minutes. An optional dose will be given when the initial examination is not conclusive, e. g. when the arterial phase is partly missed. When both examinations are done the lesions were classified using the Bosniak classification system and a comparison of both methods will be done.

ELIGIBILITY:
Inclusion Criteria:

* Finding of a complex cystic renal lesion

Exclusion Criteria:

* age < 18 y, gravity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a CT procedure.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Hohmann, MD, Principal Investigator — Department of Radiology, University Hospital Basel, University of Basel
Locations (1):
- Department of Radiology, University Hospital Basel, University of Basel, Basel, Switzerland